CLINICAL TRIAL: NCT06396143
Title: Research on Intelligent Screening and Decision-making for Neoadjuvant Therapy in Locally Advanced Gastric Cancer Based on Multi-omics Integration
Status: Recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Jian Chen, Head of Gastrointestinal Surgery, Second affiliated hospital of Zhejiang university School of Medicine, Zhejiang University
Other Study IDs: WKJ-ZJ-2310
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Locally Advanced Gastric Carcinoma
Keywords: Gastric cancer; Neoadjuvant chemotherapy; Immunotherapy; Targeted therapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Neoadjuvant chemotherapy group: a. Pathological diagnosis of gastric adenocarcinoma; b. The CT evaluation of gastric cancer is clinical stage II-IVa (≥ T3, and/or lymph node positive), with or without local tissue or organ invasion, and no distant metastasis; c. Acceptance criteria for 2-4 courses of 5-FU+platinum based neoadjuvant chemotherapy regimen. D2 gastric cancer radical surgery will be performed after the neoadjuvant treatment regimen； e. Enhanced CT images and digital images of HE stained gastroscopy biopsy sections before neoadjuvant therapy are available; f. Complete clinical diagnosis and treatment information, as well as expression information of targeted and immunotherapy related molecular markers.
- Neoadjuvant chemotherapy combined with PD1 or PDL1 group: a. Pathological diagnosis of gastric adenocarcinoma; b. The CT evaluation of gastric cancer is clinical stage II-IVa (≥ T3, and/or lymph node positive), with or without local tissue or organ invasion, and no distant metastasis; c. Acceptance criteria for a 2-4 course treatment regimen based on 5-FU+platinum neoadjuvant chemotherapy combined with anti PD-L1 therapy; d. D2 gastric cancer radical surgery was performed after the new adjuvant treatment regimen; e. Enhanced CT images and digital images of HE stained gastroscopy biopsy sections before neoadjuvant therapy are available; f. Complete clinical diagnosis and treatment information, as well as expression information of targeted and immunotherapy related molecular markers.
- Neoadjuvant chemotherapy combined with trastuzumab group: a. Pathological diagnosis of gastric adenocarcinoma; b. The CT evaluation of gastric cancer is clinical stage II-IVa (≥ T3, and/or lymph node positive), with or without local tissue or organ invasion, and no distant metastasis; c. Acceptance criteria for 2-4 courses of 5-FU+platinum neoadjuvant chemotherapy combined with trastuzumab regimen; d. D2 gastric cancer radical surgery was performed after the new adjuvant treatment regimen; e. Enhanced CT images and digital images of HE stained gastroscopy biopsy sections before neoadjuvant therapy are available; f. Complete clinical diagnosis and treatment information, as well as expression information of targeted and immunotherapy related molecular markers.

SUMMARY:
In this study, investigators utilize a radiopathomics integrated Artificial Intelligence (AI) supportive system to predict tumor response to neoadjuvant chemoradiotherapy (nCRT) before its administration for patients with locally advanced gastric cancer (LAGC). By the system, the postoperative tumor regression grade (TRG) of the participants will be identified based on the radiopathomics features extracted from the pre-nCRT Enhanced CT and biopsy images. The ability to predict TRG will be validated in this multicenter, prospective clinical study.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational clinical study for validation of a radiopathomics artificial intelligence (AI) system. Patients who have been diagnosed with gastric adenocarcinoma by pathology and defined as clinical stage II-IVa without distant metastasis by enhanced CT scan will be enrolled from the Second Affiliated Hospital of Zhejiang University, the First Affiliated Hospital of Zhejiang University, Shangyu People's Hospital of Shaoxing City and Zhejiang Cancer Institute & Hospital. All participants should adhere to a highly standardized treatment protocol, which involves receiving either 2-4 courses of standard neoadjuvant chemotherapy based on 5-FU + platinum, or 2-4 courses of neoadjuvant chemotherapy based on 5-FU + platinum combined with trastuzumab, or 2-4 courses of neoadjuvant chemotherapy based on 5-FU + platinum combined with anti-PD-L1 therapy. Following the neoadjuvant treatment protocol, participants will undergo a D2 radical gastrectomy for gastric cancer. The enhanced CT and biopsy examination should be completed before the nCRT and the images will be subjected to the manual delineation of the tumor regions of interest (ROI) by experienced radiologists and pathologists. Subsequently, the enhanced CT and biopsy images outlined will be used in the radiological pathology AI system to generate predicted responses (predicted postoperative TRG grading) for individual patients, while actual responses (confirmed postoperative TRG grading) will be diagnosed in surgical resection specimens. Through comparisons of the predicted responses and true pathologic responses, investigators calculate the prediction accuracy, specificity, sensitivity as well as the Area Under Curve (AUC) of Receiver Operating Characteristic (ROC) curves. The aim of this study is to verify the high accuracy and robustness of the radiological pathology AI system in predicting postoperative TRG grading in individuals before nCRT, which will promote further precise treatment of locally advanced cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of gastric adenocarcinoma
2. Gastric cancer CT evaluation is clinical stage II-IVa (≥ T3, and/or lymph node positive), with or without local tissue or organ invasion, and no distant metastasis.
3. Acceptance criteria for 2-4 courses of 5-FU+platinum neoadjuvant chemotherapy regimen, or 2-4 courses of 5-FU+platinum neoadjuvant chemotherapy combined with trastuzumab regimen, or 2-4 courses of 5-FU+platinum neoadjuvant chemotherapy combined with anti-PD-L1 treatment regimen.
4. D2 gastric cancer radical surgery after neoadjuvant therapy
5. Digital images of enhanced CT images and HE stained gastroscopy biopsy sections before neoadjuvant therapy are available.
6. Complete clinical diagnosis and treatment information, as well as expression information of targeted and immunotherapy related molecular markers.

Exclusion Criteria:

1. Has a history of other tumors.
2. Insufficient imaging quality of CT or biopsy slides, unable to obtain features.
3. Unable to extract molecular information related to research from organizational samples.
4. Interruption of neoadjuvant therapy course for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population in the study is LAGC patients who plan to receive standard neoadjuvant concurrent chemotherapy or combination immunotherapy and targeted therapy, but the tumor pathological response is unknown.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The area under curve (AUC) of Receiver Operating Characteristic (ROC) curves of the radiopathomics artificial intelligence model | baseline
  Calculate the area under the receiver operating characteristic (ROC) curve (AUC) of the artificial intelligence model for radiomics to predict the postoperative pathological TRG grading index in LAGC patients treated with nCRT.

SECONDARY OUTCOMES:
The specificity of the radiopathomics artificial intelligence model | baseline
  the specificity of artificial intelligence models for radiomics in predicting postoperative TRG grading in LAGC patients treated with nCRT.
The sensitivity of the radiopathomics artificial intelligence model | baseline
  The sensitivity of artificial intelligence models for radiomics in predicting postoperative TRG grading in LAGC patients treated with nCRT.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Gastrointestinal Department of First Affiliated Hospital of Zhejiang University, Hanzhou, Zhejiang
  - Gastrointestinal Department of Second Affiliated Hospital of Zhejiang University, Hanzhou, Zhejiang
  - Gastrointestinal Department of Zhejiang Cancer Hospital, Hanzhou, Zhejiang
  - Shaoxing Shangyu People's Hospital, Shaoxing, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feng L, Liu Z, Li C, Li Z, Lou X, Shao L, Wang Y, Huang Y, Chen H, Pang X, Liu S, He F, Zheng J, Meng X, Xie P, Yang G, Ding Y, Wei M, Yun J, Hung MC, Zhou W, Wahl DR, Lan P, Tian J, Wan X. Development and validation of a radiopathomics model to predict pathological complete response to neoadjuvant chemoradiotherapy in locally advanced rectal cancer: a multicentre observational study. Lancet Digit Health. 2022 Jan;4(1):e8-e17. doi: 10.1016/S2589-7500(21)00215-6. PMID 34952679